CLINICAL TRIAL: NCT05011773
Title: Manipulating and Optimising Brain Rhythms for Enhancement of Sleep
Acronym: MORPHEUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Surrey Sleep Research Centre, Surrey, UK (Unknown); Mayo Clinic (Other); University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 20/PR/0409
Record Dates: First submitted 2021-08-04; First posted 2021-08-18 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-10

CONDITIONS: Parkinson Disease; MSA - Multiple System Atrophy; Chronic Pain; Epilepsy
Keywords: sleep; Electroencephalography; Deep brain stimulation
MeSH Terms: conditions — Parkinson Disease; Shy-Drager Syndrome; Chronic Pain; Epilepsy | interventions — Deep Brain Stimulation

STUDY DESIGN:
Intervention Model Description: Evaluation of symptomatology "on" and "off" deep brain stimulation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Deep brain stimulation (Experimental): All patients have already undergone deep brain stimulation. Results compared "on" and "off" stimulation.
  Interventions: Device: Deep brain stimulation

INTERVENTIONS:
Device: Deep brain stimulation — Electrical pulses from implanted generator that has already been implanted for therapeutic reasons

SUMMARY:
Treatment of sleep disturbances is mainly attempted through drug administration. However, certain drugs are associated with unwanted side effects or residual effects upon awakening (e.g. sleepiness, ataxia) which can increase the risks of falls and fractures. In addition, there can be systemic consequences of long-term use. An alternative method of manipulating sleep is by stimulating the brain to influence the electroencephalogram (EEG). To date, there have been mixed results from stimulating superficial areas of the brain and, as far as we know, there has been no systematic attempt to influence deep brain activity.

Many patients suffering from movement disorders, such as Parkinson's Disease (PD) and Multiple Systems Atrophy (MSA), also have disrupted sleep. Currently, at stages where drug treatment no longer offers adequate control of their motor symptoms, these patients are implanted with a deep brain stimulation system. This involves depth electrodes which deliver constant pulse stimulation to the targeted area. A similar system is used in patients with severe epilepsy, as well as some patients with chronic pain.

The aim of this feasibility study is to investigate whether we can improve sleep quality in patients with deep brain stimulators by delivering targeted stimulation patterns during specific stages of sleep. We will only use stimulation frequencies that have been proven to be safe for patients and frequently used for clinical treatment of their disorder. We will examine the structure and quality of sleep as well as how alert patients are when they wake up, while also monitoring physiological markers such as heart rate and blood pressure. Upon awakening, we will ask the patients to provide their subjective opinion of their sleep and complete some simple tests to see how alert they are compared to baseline condition which would be either stimulation at the standard clinical setting or no stimulation.

We hope that our study will open new ways of optimising sleep without the use of drugs, in patients who are implanted with depth electrodes. We also believe that our findings will broaden the understanding of how the activity of deep brain areas influences sleep and alertness.

DETAILED DESCRIPTION:
This is a feasibility study that will take place in two UK sites: the John Radcliffe Hospital (Oxford) and the Surrey Sleep Research Centre, University of Surrey. The identification, consent and screening of patients will take place in Oxford, and the sleep assessments will take place in Surrey. A parallel study will also be conducted at US sites (Mayo Clinic, Rochester MA, and UCSF, CA) under the same funding but this will be reviewed by their local IRB. De-identified data may be shared between sites for analyses purposes. This will be done securely in an encrypted fashion while participants will be made fully aware of this.

Participants will be identified during their routine clinic visits with the Functional Neurosurgery team (John Radcliffe Hospital) and invited to participate in the study. Screening of interested potential participants will take into account pre-operative assessment data. Testing will ensue (within a variable period from screening, but within the aforementioned study timeline), over two visits to the Surrey Sleep Research Centre, each consisting of two nights. The maximum duration between consent and first study visit will be three months, while there will be a minimum of two weeks between each study visit to allow for preliminary analyses. Informed consent and baseline sleep recordings will be obtained over the first night of the first visit to Surrey, with the remaining nights consisting of stimulation trials. Questionnaires, daytime vigilance testing, autonomic parameters and cortisol levels will be collected. No long-term follow-up is planned at this stage.

With regards to data collection processes, the population of patients visiting the Surrey site will have already been implanted with a DBS system (such as an Activa PC/PC+S (Medtronic) or an Abbot/St Jude device). The investigators will leverage rules from the current AASM guidelines, technologies and methods for manual and automated sleep scoring using standard scalp polysomnography as well as novel methods we previously developed for sleep scoring using intracranial electrophysiology. To avoid contamination of the electrophysiology monitoring amplifiers by the stimulation protocol, a combination of bipolar stimulation and sampling-stimulate rate interactions will be used. For example, we will apply know-how from the Activa PC+S work to place any residual artefacts into bands of little physiological interest (DC, 50/60Hz, etc.). A preliminary assessment of amplifier performance will provide assurance that we will be able to maintain sleep staging accuracy over the course of our experiments.

For perturbations, the CE-marked clinician programmer will be used (especially at the open-loop stage) or a research variant thereof. In this study, high-frequency (HF) is specified at a stimulation range from 41Hz to 250Hz, while low frequency (LF) will be defined as 2-40Hz. All perturbations will be within the clinical range used and approved for DBS patients. A combination of subjective and objective measurements of sleep quality and efficiency to measure the impact of any sleep perturbations will be used.

The following objective metrics will be derived from visual/manual polysomnography (gold standard) & automated algorithm sleep staging:

1. Total sleep time.
2. Number of sleep cycles (switches of non-rapid eye movement (NREM) and rapid eye movement (REM) sleep).
3. Initial sleep and REM latencies (Time from beginning of study to the first stage of sleep, and from beginning of sleep to first REM sleep onset).
4. Duration of N1, N2, N3, and REM stages, and the duration of NREM (sum of N1,N2,N3)stages.
5. Sleep efficiency (100*total sleep time/time in bed).
6. Number of awakenings during night, including arousals per hour and duration of time spent awake after initial sleep onset (i.e., wake after sleep onset time)
7. Apnoea-hypopnea and respiratory disturbance indices (the frequency of stop or reduced breathing episodes, and respiratory arousals per hour)
8. Periodic limb movement indices (the frequency of periodic leg movements of sleep per hour)
9. Measures of arousal during sleep

   1. behavioural macrostate observations such as eye opening or blinking that can be assessed in video recordings
   2. microarousal observations defined exclusively by cortical fast frequency shifts (ie, >14 Hz rhythms) lasting 3 seconds or longer, with or without added autonomic measures of tachycardia.
   3. Spectral composition of the sleep stage specific EEG over the 0.25-32 Hz frequency range Salivary samples to characterize awakening levels of cortisol will be obtained in the Surrey Sleep Research Centre at the end of each night.

Questionnaires will be administered to patients such as those listed below (not all necessary):

Upon enrolment/prior to the participant's visit:

* Pittsburgh Sleep Quality Index (PSQI) (Buysse et al 1989)
* Movement Disorder Society-Sponsored Revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS) (last amendment 2019, original article Goetz et al 2008)
* Parkinson's Disease Sleep Scale (PDSS) (Trenkwalder et al. 2011)
* Patient sleep diary (bedtime, awakening time, arousals/sleep disturbances, perceived sleep quality)

During the visits to the Surrey Sleep Research Centre:

* Karolinska Sleepiness Scale (KSS) (Akerstedt and Gillberg, 1990)
* Samn Perelli Fatigue Scale (Samn and Perelli, 1982)
* Profile of Mood States Scale (POMS) (McNair, Lorr and Doppleman, 1971)

With regards to collecting data relevant to cognitive performance, we will focus on assessments of sleep inertia as measured by performance characteristics assessed by tasks listed below:

* Digit Symbol Substitution Test (DSST) (as in Boyle et al. 2012)
* Psychomotor Vigilance Task (PVT) (as in Santhi et al. 2013)
* N-back task (Santhi et al. 2013)
* Karolinska Drowsiness Test (KDT) (Akerstedt and Gillbert, 1990)

ELIGIBILITY:
Inclusion Criteria:

* Either already implanted with DBS electrodes or undergoing DBS implantation in one of the defined nuclei of interest (for Surrey or Rochester: STN, PPN, Hypothalamus, PAG/PVG - for the Mayo clinic, may use hippocampus or ANT) for standard clinical care during the period of the study
* Male or female, aged 18 to 85
* Be willing and able to give written and oral informed consent
* Ability to complete all required study procedures including travelling to the Sleep Centre and staying overnight
* By the time of the first visit to Surrey, participants should have already had their stimulation settings programmed by the Functional Neurosurgery team and have been stable on the settings for at least two weeks, as per their routine clinical care.
* For patients with chronic pain, they should be stable on their current medication and settings

Exclusion Criteria:

* Cognitive impairment (judged by the clinician taking consent as not having sufficient mental capacity to understand the study and its requirements). This is including anyone who, in the opinion of the clinician taking consent is unlikely to retain sufficient mental capacity for the duration of their involvement in the study.
* Patients with any other medical condition that would interfere with study conduct or make it unsafe for them to participate. Such conditions may be poorly controlled diabetes, poorly controlled/end stage heart disease, renal failure as well as recurrent, uncontrolled seizures or epilepsy.
* Participants who have started new medication or changed doses 3 weeks prior to a study visit may not be eligible as deemed by the PI of the study.
* Patients on medication that can affect the study results (such as hypnotics - benzodiazepines and analogues), at the discretion of the PI.
* Patients currently taking ketamine
* Alcohol intake exceeding 28 units per week.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2021-08-03 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Sleep stages | 4 nights total (2 visits of 2 nights with DBS ON and OFF during each visit). Each night is defined as the period between 2300hrs and 0700 hrs in a windowless, temperature controlled sleep laboratory
  Sleep staging will assessed using gold standard sleep polysomnography (Video EEG, EOG, ECG). Sleep stage classification will be assessed by an expert sleep neurophysiologist using standard AASM and other criteria. DBS ON and night and DBS OFF night will be compared to look for the differences in sleep architecture such as total sleep time and duration in sleep phase (N1-3, REM, non-REM and wakefulness)
Sleep inertia | 4 nights total (2 visits of 2 nights - same period as outcome 1)
  Differences in sleep inertia after DBS ON vs DBS OFF night will be compared using the sleep inertia scale (questionnaire)

SECONDARY OUTCOMES:
Control of sleep | 4 nights total (2 visits of 2 nights - same period as outcome 1)
  To assess the possibility of controlling sleep depth and sleep wake transitions by DBS. This will be assessed by comparing stages of sleep to awakenings and time spent in transition between sleep stages (comparing DBS ON to DBS OFF)

OTHER OUTCOMES:
Heart rate variability | 4 nights total (2 visits of 2 nights - same period as outcome 1)
  Overnight continuous measurements during study. Heart rate variability will be calculated from continuous ECG using standard techniques such as power spectral analysis
Blood pressure | 4 nights total (2 visits of 2 nights - same period as outcome 1)
  Measured using ambulatory non-invasive cuff method immediately prior to sleep and upon waking. SBP and DBP will be measured and and compared between DBS ON and OFF
Salivary cortisol levels | 4 nights total (2 visits of 2 nights - same period as outcome 1)
  Measured upon wakening and 30/60/90 mins after wakening each day during study. Levels will be compared between periods after DBS ON and DBS OFF.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander L Green, FRCS(SN), Principal Investigator — Oxford University Hospitals NHS Trust
Locations (1):
- John Radcliffe Hospital, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
We are recruiting only 20 patients, so sharing IPD even anonymised, may be identifiable. Decision will be taken when this can be definitively elucidated.